CLINICAL TRIAL: NCT06773494
Title: Long-term Clinical and Radiographic Evidence of Alleviation of Preoperative Chronic Sinusitis After Open Sinus Allogeneic Bone Augmentation Surgery: A Retrospective Observational Study
Brief Title: Clinical and Radiographic Evidence of Alleviation of Preoperative Chronic Sinusitis After Open Sinus Allogeneic Bone Augmentation Surgery: A Retrospective Observational Study
Status: Completed | Type: Observational
Sponsor: Misr International University (Other)
Collaborators: Suez Canal University (Other)
Responsible Party: Principal Investigator, Hebatallah Abdo's Elsaid Mattar, Assistant Lecturer, Misr International University
Other Study IDs: 2024/518
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Chronic Sinusitis; Open Sinus Elevation
Keywords: open sinus elevation; lateral window; dental implants; chronic sinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the impact of open sinus elevation technique on chronic sinusitis when combined with simultaneous dental implant placement. A retrospective analysis of patients with chronic sinusitis who underwent sinus elevation and dental implant procedures was performed. Radiographic images were analyzed preoperatively and postoperatively to assess the fluid levels in the sinuses. Clinical evaluation through a questionnaire tabulated by an ENT specialist was done for all patients. The results showed the following: Preoperative radiographs showed varying fluid levels in the sinuses. Postoperative results demonstrated that fluid levels were either entirely eliminated or significantly reduced in all cases. Therefore, it can be concluded that sinus elevation procedures, when performed concurrently with dental implants, can alleviate chronic sinusitis symptoms as evidenced by reduced fluid levels in the sinus cavities.

DETAILED DESCRIPTION:
Introduction Implant placement in the posterior maxilla may be a dilemma. Factors complicating the treatment may be anatomical landmarks, type of bone, residual bone height, limited accessibility, maxillary sinus pneumatization as well as sinus pathologies such as chronic or acute sinusitis (1,2).

When vertical bone in the posterior maxilla is compromised due to maxillary sinus pneumatization several protocols were advocated to overcome this occurrence, such as the placement of short implants (3), 2nd premolar occlusion (4), or maxillary sinus elevation (5). Sinus elevation was introduced in 1980 when Boyne and James presented the lateral window approach as a modification of the Caldwell- Luc technique; access to lift the sinus floor is performed by a window through the lateral wall of the sinus (6). This technique was proven to be effective and successful for sinus elevation, even up to 12 mm in cases of severely atrophic ridge (7). It was later divided into three techniques according to the lateral wall preparation: hinge, elevated, and complete (8).

The high position of the Maxillary Sinus Ostium (MSO) led to the fact that drainage of the sinus is always against the gravitational force, an important factor that may lead to fluid precipitation inside the sinus and needs to be considered when dealing with maxillary sinusitis (9).

The presence of pre-operative sinus pathologies, including chronic and acute sinusitis may complicate the treatment of open sinus elevation as they may affect the integrity of the Schneiderian membrane at the time of open sinus elevation (10). Not only so, but they may also increase the risk of post-operative sinusitis (11).

However, a research gap exists in this aspect since a systematic review published in 2021 negated that suggestion and mentioned that mucosal thickenings of the Schneiderian membrane and/ or chronic sinusitis are not likely to pause extra risk factors in terms of sinus augmentation (12).

Patients and Methods

Patient Selection:

The current research was performed on 36 sinuses selected from patients in Oral and Maxillofacial outpatients' clinics at the Faculty of Dentistry, Suez Canal University, who underwent sinus lifting procedures to increase alveolar ridge height for simultaneous implant placement. The study was planned as a comparative retrospective study under the World Medical Association Declaration of Helsinki. All clinical and radiographic data will be acquired through the screening of saved patients' files, radiographs and a patient filled questionnaire. The selected patients' records fulfilled selective criteria.

Inclusion Criteria:

1. Males and females ≥ 18 years of age.
2. ASA I and ASA II.
3. Patients having partial edentulism in the posterior region of the maxilla.
4. Edentulous sites consist of native non augmented bone.
5. Horizontal ridge dimension minimum of 5mm
6. The vertical ridge dimension 4-7 mm.
7. Bone quality of D2 or D3.
8. Enough inter-arch distance.
9. The presence of one-year postoperative radiograph CBCT.
10. Presence of postoperative follow up clinical data.

Exclusion Criteria:

1. Patients with active acute infection or residual lesion related to the edentulous sites.
2. Acute maxillary sinus pathosis
3. A remaining root dislodged in the Maxillary sinus.
4. Patients that lack a stable occlusion or have parafunctional habits.
5. Patients with poor oral hygiene who are not amenable to motivation and improvement.
6. Smokers who smoke more than 10 cigarettes a day.
7. Pregnant or lactating mothers.
8. Alcohol and drug abuse.
9. Treatment with radiation therapy in the craniofacial region within the previous 12 months.

Surgical protocol:

All the surgical procedures were performed by the same surgeon using standardized techniques under aseptic conditions. Open sinus elevation was done with simultaneous implant placement with allogenic bone graft. The follow up period for all patients was one year.

Outcomes assessment:

Clinical outcomes:

Clinical examination was done by an ENT specialist, where the patient filled a questionnaire (formulated by the ENT specialist) which was used to determine the presence or absence of symptoms of chronic sinusitis.

Radiographic outcomes:

All subjects were evaluated for presence or absence of chronic sinusitis in the preoperative CBCT and one-year follow up CBCT. Fusion module was used to accurately compare both CBCTs by superimposing the postoperative CBCT on the preoperative CBCT.

Chronic sinusitis is identified as the presence of thickening of Schneiderian membrane ≥ 2 mm, mucosal cyst, polyp, or fluid level (13).

Statistical Plan:

Sample size calculation:

This power analysis used bone height gain as the primary outcome. The effect size f = (3.2349048) was calculated based upon the results of Hammuda & ghoneim 2021 (13) and assuming that the standard deviation within each group = 0.8, using alpha level of 5% and Beta level of 20% i.e. power = 80%. The minimum estimated sample size was 8 samples per group. Sample size calculation was done using G*Power version 3.1.9.2

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females ≥ 18 years of age. 2. ASA I and ASA II. 3. Patients having partial edentulism in the posterior region of the maxilla. 4. Edentulous sites consist of native non augmented bone. 5. Horizontal ridge dimension minimum of 5mm 6. The vertical ridge dimension 4-7 mm. 7. Bone quality of D2 or D3. 8. Enough inter-arch distance. 9. The presence of one-year postoperative radiograph CBCT. 10. Presence of postoperative follow up clinical data.

Exclusion Criteria:

* 1. Patients with active acute infection or residual lesion related to the edentulous sites.

  2. Acute maxillary sinus pathosis 3. A remaining root dislodged in the Maxillary sinus. 4. Patients that lack a stable occlusion or have parafunctional habits. 5. Patients with poor oral hygiene who are not amenable to motivation and improvement.

  6. Smokers who smoke more than 10 cigarettes a day. 7. Pregnant or lactating mothers. 8. Alcohol and drug abuse. 9. Treatment with radiation therapy in the craniofacial region within the previous 12 months.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The current research was performed on 36 sinuses selected from patients in Oral and Maxillofacial outpatients' clinics at the Faculty of Dentistry, Suez Canal University, who underwent sinus lifting procedures to increase alveolar ridge height for simultaneous implant placement. The study was planned as a comparative retrospective study under the World Medical Association Declaration of Helsinki. All clinical and radiographic data will be acquired through the screening of saved patients' files, radiographs and a patient filled questionnaire. The selected patients' records fulfilled selective criteria.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Radiographic outcome | 1 year
  All subjects were evaluated for presence or absence of chronic sinusitis in the preoperative CBCT and one-year follow up CBCT. Fusion module was used to accurately compare both CBCTs by superimposing the postoperative CBCT on the preoperative CBCT.
  Chronic sinusitis is identified as the presence of thickening of Schneiderian membrane ≥ 2 mm, mucosal cyst, polyp, or fluid level.

SECONDARY OUTCOMES:
Clinical outcome | 1 year
  Clinical examination was done by an ENT specialist, where the patient filled a questionnaire (formulated by the ENT specialist) which was used to determine the presence or absence of symptoms of chronic sinusitis.

CONTACTS AND LOCATIONS:
Overall Officials: Hebatullah A Mattar, Assistant Lecturer, Principal Investigator — Misr International University; Wael A Hussein, Assistant Lecturer, Study Director — Misr International University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided